CLINICAL TRIAL: NCT06527469
Title: Intensive Pediatric Group Intervention in a Curricularly-embedded Pro-bono Clinic
Brief Title: Intensive Pediatric Group Intervention
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jamie Hall, Associate Teaching Professor, Principal Investigator, University of Missouri-Columbia
Other Study IDs: 2113446
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy
Keywords: physical therapy; power training; strength training; pediatrics; gait training; group therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PhysZou emPOWER: Strength, power, and gait-based intervention for kids with cerebral palsy is embedded within a curricular pro-bono student physical therapy clinic. The group will meet for 2 hours, 2 times per week for 15 weeks.
  Interventions: Other: PhysZou emPOWER: a strength, power, and gait intervention group physical therapy program for children with CP

INTERVENTIONS:
Other: PhysZou emPOWER: a strength, power, and gait intervention group physical therapy program for children with CP — Each session will include a 10-minute game-based warm-up, 45 minutes of gait interventions to include treadmill and overground walking as well as other aerobic activities, 45 minutes of resistance training (power and strength training as appropriate for their individual goals), and a 10-minute cool-down incorporating yoga and breathing activities. To ensure participants are exercising at the appropriate level of intensity, 1 repetition maximum measures will be used to determine the appropriate levels of resistance and heart rate monitors will be worn.

SUMMARY:
The purpose of the Mizzou emPOWER program is to meet the curricular needs of entry-level doctorate of physical therapy students by providing them the real-world experience of implementing recent evidence surrounding physical therapy dosing for children with cerebral palsy (CP) for power, strength, and gait interventions while meeting an unmet community need.

DETAILED DESCRIPTION:
Beginning in Fall 2024, the investigators will recruit 6 children with CP, Gross Motor Function Classification System Levels I-III, ages 7-17 years old, to participate in the program. Two students will be assigned to each participant, rotating every 4 weeks due to the structure of the pro-bono clinic. A total of 3 faculty members will supervise. The group will meet for 2 hours, 2 times per week for 15 weeks. Each session will include a 10-minute game-based warm-up, 45 minutes of gait interventions to include treadmill and overground walking as well as other aerobic activities, 45 minutes of resistance training (power and strength training as appropriate for their individual goals), and a 10-minute cool-down incorporating yoga and breathing activities. Participant assessments will be completed during the first week, 7th week, and 15th week. Other programmatic assessments will include students' written reflections on their experiences providing this program, caregiver satisfaction surveys, and participant and caregiver interviews.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory children 7-17 years old, children who are participating in emPOWER program
* GMFCS Levels I-III
* Able to follow 2-3 step directions
* English Speaking

Exclusion Criteria:

* Orthopedic surgery in the past year
* Significant visual impairment
* Significant hearing impairment

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Ambulatory children aged 7-17 years old with Cerebral Palsy (GMFMCS Levels I-III), participating in PhysZou emPOWER program.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
1 Repetition Maximum (1-RM) Testing | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Particpants will complete strength testing of hip/knee extensors and plantarflexor muscle groups using a leg press, using 1 Rep max testing protocols, as outlined in Pontiff and moreau, 2022. (PMID 35960137)
10 meter walk test | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Walking speed test of 10 meter distance, completed in both conditions of self selected speed and fast gait speed
Keiser Leg Press | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Assessment of lower extremity power
Timed up and Down Stairs | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Functional measure of how quickly child can climb up and down 1 flight of stairs
30 second sit to stands | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  This is a clinical assessment of lower extremity strength, in which investigators count the number of repetitions of sit to stands completed in 30 seconds.
30 second half kneel to stand | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  This is a clinical assessment of lower extremity strength, in which investigators count the number of repetitions of half kneel to stand complete correctly in a 30 second time period.
Lateral Step Ups | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  This is a clinical assessment of lower extremity strength, in which investigators count the number of repetitions of lateral step ups completed in 30 seconds on a standard size 6 inch step.
Gross Motor Function Measure-88 (GMFM-88) | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  This is a criterion referenced measure of gross motor function and is valid and reliable for children with cerebral palsy. It evaluates motor skills that are typical for normal development. Dimensions D and E will be utilized, as these 2 sections assess the overall gross motor function in direct relation to standing, walking, running, and jumping.
Canadian Occupational Performance Measure | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Evidence-based outcome measure designed to capture a client's self-perception of performance in goals they determine before intervention. The measurement focuses on self-care, leisure activities, and productivity. The participant rates their performance and their satisfaction with their performance on a scale from 1-10, with 1 indicating poor performance and low satisfaction, while 10 indicates very good performance and high satisfaction.
Standing balance with eyes closed standing on firm surface | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Participants will stand on a force plate with eyes closed. Postural control information is obtained from the investigators and the force plate tracks the center of pressure of the participant.
Standing balance with eyes closed standing on firm surface | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Joint kinematics (movement strategies) obtained while eyes closed standing on firm surface
Walking- single task | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Walking speed is obtained form spatial sensor
Walking- single task | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Stride length obtained from spatial sensor
Walking- cognitive dual task | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  speed of walking will be obtained from spatial sensor while completing appropriate/salient cognitive dual task
Walking- cognitive dual task | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  stride length will be obtained from spatial sensor while completing appropriate/salient cognitive dual task
5 Times sit to stand test | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  time to complete and knee joint kinematics obtained from spatial sensor
Step down | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  knee joint kinematics obtained from spatial sensor while the participant steps down from a 6 inch curb step
Jumping | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Production of power will be obtained from force plate and spatial sensor
Jumping | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  Assessment of knee joint kinematics during jumping will be obtained from force plate and spatial sensor
Reaction time | Before PT intervention begins (week 1), midpoint of program (Week 7), and last week of program (week 15).
  measurement of upper extremity reaching reaction

SECONDARY OUTCOMES:
Perspectives of children and caregivers | Completion of program (Week 15)
  Semi-structured interviews will provide researchers with the perspective of the children and caregivers who participated in this novel program.
Perspectives of children and caregivers | Completion of program (Week 15)
  Open ended surveys will provide researchers with the perspective of the children and caregivers who participated in this novel program.
Perspectives of Doctor of Physical Therapy Students | Completion of program (week 15)
  Open ended surveys will provide researchers and faculty with the perspective of the learning opportunity from the students

CONTACTS AND LOCATIONS:
Locations (1):
- PhysZou-University of Missouri Department of Physical Therapy, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambuehl M, van Hedel HJA, Labruyere R. Pediatric Rehabilitation Therapies Differ in Intensity: A Pilot Study to Highlight the Implications for Dose-Response Relationships. Am J Phys Med Rehabil. 2020 Mar;99(3):224-232. doi: 10.1097/PHM.0000000000001323. PMID 31592876
- [Background] Bjornson KF, Moreau N, Bodkin AW. Short-burst interval treadmill training walking capacity and performance in cerebral palsy: a pilot study. Dev Neurorehabil. 2019 Feb;22(2):126-133. doi: 10.1080/17518423.2018.1462270. Epub 2018 Apr 16. PMID 29658831
- [Background] Hedgecock JB, Harris NM, Rapport MJ. Changing Practice: Clinical Application of Resistance Training Evidence for Children With Cerebral Palsy. Pediatr Phys Ther. 2023 Jul 1;35(3):367-376. doi: 10.1097/PEP.0000000000001023. PMID 37289202
- [Background] Oudenhoven LM, van Vulpen LF, Dallmeijer AJ, de Groot S, Buizer AI, van der Krogt MM. Effects of functional power training on gait kinematics in children with cerebral palsy. Gait Posture. 2019 Sep;73:168-172. doi: 10.1016/j.gaitpost.2019.06.023. Epub 2019 Jul 16. PMID 31344605
- [Background] van Vulpen LF, de Groot S, Rameckers E, Becher JG, Dallmeijer AJ. Improved Walking Capacity and Muscle Strength After Functional Power-Training in Young Children With Cerebral Palsy. Neurorehabil Neural Repair. 2017 Sep;31(9):827-841. doi: 10.1177/1545968317723750. Epub 2017 Aug 8. PMID 28786309
- [Background] Pontiff M, Moreau NG. Safety and Feasibility of 1-Repetition Maximum (1-RM) Testing in Children and Adolescents With Bilateral Spastic Cerebral Palsy. Pediatr Phys Ther. 2022 Oct 1;34(4):472-478. doi: 10.1097/PEP.0000000000000941. Epub 2022 Aug 12. PMID 35960137